CLINICAL TRIAL: NCT00256802
Title: The Diameter of the Middle Cerebral Artery Measured With Magnetic Resonance Angiography (MRA) Under Provocation With Glyceryl Trinitrate in Healthy Volunteers.
Brief Title: The Diameter of the Middle Cerebral Artery Measured With Magnetic Resonance Angiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: MRA-GTN2004
Record Dates: First submitted 2005-11-21; First posted 2005-11-22 (Estimated); Last update posted 2009-04-01 (Estimated); Status verified 2004-05

CONDITIONS: Headache; Migraine; MR-Angiography; Healthy Volunteers; GTN; Middle Cerebral Artery
Keywords: Headache; migraine; MR-angiography; healthy volunteers; GTN; Middle cerebral artery
MeSH Terms: conditions — Headache; Migraine Disorders | interventions — Magnetic Resonance Angiography

INTERVENTIONS:
Device: MR-angiography, GTN

SUMMARY:
To examine the ability of MRA to measure the effect of GTN on the intra-cranial vascular response during the GTN-induced headache in healthy volunteers.

DETAILED DESCRIPTION:
The only intra cranial structures innervated by sensory nerves, and therefore a possible source of the headpain are the meninges and the large intracerebral arteries. The dilatation of the cerebral vessels may not be the origin of the head pain per se, but measurements of the intra cerebral vascular bed in the past has proven valuable in the migraine-research, and has helped elucidate the basis for the migraine aura (Olesen, Friberg et al. 1990). The effects of different signal molecules on the intra cerebral vasculature continue to be an important field in the migraine research, in the search for possible pain causing signaling molecules.

Therefore we have set up at study to examine if MR-Angiography (MRA) can be used for monitoring of the vascular response after challenge with the known vasodilator GTN. This drug was chosen because it is well characterized and a large body of evidence from earlier studies could serve as background data (Thomsen 1997).

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* history of migraine or any other type of primary headaches; any kind of daily medication (including prophylactic headache therapy but not oral contraceptives); excessive use of analgesics (corresponding to >2 g aspirin/day), pregnancy and all known contraindications for MR-examinations incl. claustrophobia.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12
Dates: Start 2004-06; Study Completion 2005-01

PRIMARY OUTCOMES:
The primary endpoints were the difference between the area under the curve of the MCA area and the difference between the area under the curve of the diameter of the MCA on an active day and on a placebo day recorded over 60 mins.

SECONDARY OUTCOMES:
The secondary endpoints were difference in the area under the curve for the relative changes in area in percent deviation from baseline, and the difference in headache response.

CONTACTS AND LOCATIONS:
Overall Officials: Jakob Møller Hansen, MD, Study Chair — Danish Headache Center

REFERENCES:
- See also: The homepage of the Danish headache center, Glostrup, Copenhagen, Denmark — http://www.glostruphospital.dk/danishheadachecenter/menu